CLINICAL TRIAL: NCT03263507
Title: A Double-Blind, Placebo-Controlled, Dose-Escalation Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ISIS 721744, an Antisense Oligonucleotide Inhibitor of PKK, Administered Subcutaneously to Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Donidalorsen (IONIS-PKK-LRx) Administered Subcutaneously to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 721744-CS1
Record Dates: First submitted 2017-08-17; First posted 2017-08-28 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Healthy Volunteers
Keywords: IONIS PKK-LRx
MeSH Terms: interventions — donidalorsen; IONIS-PKK-LRx

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Donidalorsen (Experimental): Ascending single and multiple doses of Donidalorsen administered subcutaneously
  Interventions: Drug: Donidalorsen
- Placebo (sterile saline 0.9%) (Placebo Comparator): Calculated volume to match active comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Saline .9%
  Arms: Placebo (sterile saline 0.9%)
Drug: Donidalorsen — Donidalorsen administered subcutaneously
  Other Names: ISIS 721744; IONIS-PKK-LRx
  Arms: Donidalorsen

SUMMARY:
The purpose is to assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Donidalorsen administered subcutaneously to Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent and be able to comply with all study requirements
* Healthy males or females aged 18-65 inclusive at the time of Informed Consent
* Females must be non-pregnant and non-lactating, and either surgically sterile or post- menopausal
* Males must be surgically sterile, abstinent or using an acceptable contraceptive method
* BMI <35 kg/m2

Exclusion Criteria:

* Clinically-significant abnormalities in medical history including acute coronary syndrome, major surgery within 3 months of Screening, planned surgery that would occur during the study or physical examination or other screening results such as ECGs at Screening
* Clinically significant hematologic, chemistry, and urine abnormalities
* Treatment with another Study Drug, biological agent, or device within 4 weeks of Screening
* History of bleeding diathesis or coagulopathy
* Smoking >10 cigarettes per day
* Considered unsuitable for inclusion by the Principal Investigator
* Current use of concomitant medications (including herbal or OTC medications) unless approved by Sponsor Medical Monitor
* Known history or positive test for HIV, hepatitis C or chronic hepatitis B
* Blood donation within 30 days of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events that are related to treatment with Donidalorsen | Up to 176 days
  The safety and tolerability of multiple doses of Donidalorsen will be assessed by determining the incidence, severity, and dose relationship of adverse events that are related to treatment with Donidalorsen.
Peak plasma Concentration (Cmax) of Donidalorsen | Up to 176 days
  Maximum Donidalorsen plasma concentration, Cmax (ug/mL) will be assessed following SC administration
Time to peak plasma Concentration (Tmax) of Donidalorsen | Up to 176 days
  Time to peak Donidalorsen plasma concentration, Tmax (hours) will be assessed following SC administration
Effects of Donidalorsen on plasma PKK concentration | Up to 176 days
  Effects of Donidalorsen on plasma PKK concentration after multiple doses of Donidalorsen compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Ionis Investigative Site, Toronto, Ontario, Canada